CLINICAL TRIAL: NCT03759080
Title: Mental Practice Versus Proprioceptive Neuromuscular Facilitation on Strength of Upper Limb
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to sample problem
Sponsor: Wafaa Mahmoud Amin (Other Government)
Responsible Party: Sponsor-Investigator, Wafaa Mahmoud Amin, Principal Investigator, University of Jazan
Organization: University of Jazan (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2265749560
Record Dates: First submitted 2018-11-21; First posted 2018-11-29 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: there are two arms :1. proprioceptive neuromuscular facilitation (PNF) group ,2 mental practice (MP) group.
  PNF group: 30 individuals, these subjects received PNF training. PNFMP: 30 individuals, these subjects receivedMP. training program has been administered for every group for 12 sessions over 4 weeks with 3 x 45 min training sessions per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention of PNF (Active Comparator): PNF group: 30 individuals, these subjects received proprioceptive neuromuscular facilitation training.
  Interventions: Procedure: proprioceptive neuromuscular facilitation
- MP (Experimental): PNFMP group:30 individuals, these subjects received mental practice.
  Interventions: Procedure: mental practice

INTERVENTIONS:
Procedure: mental practice — training of mental practice to do the pattern of proprioceptive neuromuscular facilitation
  Other Names: MP
  Arms: MP
Procedure: proprioceptive neuromuscular facilitation — upper limb Pattern: Flexion -Abduction- External rotation
  Other Names: PNF
  Arms: intervention of PNF

SUMMARY:
The effects of mental practice combined with proprioceptive neuromuscular facilitation on muscle strength of upper limb were measured in 60 healthy students Subjects were randomly assigned to either proprioceptive neuromuscular facilitation (PNF) group or mental practice (MP) group. PNF group: 30 individuals, these subjects received only PNF training. MP: 30 individuals, these subjects received mental practice.

DETAILED DESCRIPTION:
The effects of mental practice on muscle strength of upper limb were measured in 60 healthy female students with right dominant hand,. Their age ranged from17 to 23 years old. Subjects were randomly assigned to either proprioceptive neuromuscular facilitation (PNF) group or mental practice (MP) group. PNF group: 30 individuals, these subjects received only PNF training. MP: 30 individuals, these subjects received MP. training program has been administered for every group for 12 sessions over 4 weeks with 3 x 45 min training sessions per week. Pre-post test design was used. EMG device was used to measure the electrical activity of muscles. Measurements conducted at pre-intervention, during intervention and post-intervention testing with 20 days.

ELIGIBILITY:
Inclusion Criteria:

1.Absence of a prior injury of arm

Exclusion Criteria:

1.History of a neurological disease.

Ages: 17 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-08-20 (Estimated)

PRIMARY OUTCOMES:
Strength Evaluation of coracobrachialis Muscle | 2 minutes.
  Electromyography device was used to measure the electrical activity of muscle.
Strength Evaluation of teres minor muscle | 2 minutes.
  Electromyography device was used to measure the electrical activity of muscle.
Strength Evaluation of Brachialis muscle | 2 minutes.
  Electromyography device was used to measure the electrical activity of muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
there is no plan made